CLINICAL TRIAL: NCT00717834
Title: A Blinded Phase 1/2 Dose Escalation Study to Assess Safety and Immunogenicity and Investigate the Optimal Dose Level of a Formalin-Treated, UV-Inactivated, Vero Cell-Derived Ross River Virus (RRV) Vaccine in Healthy Volunteers Aged 18 to 40 Years
Brief Title: Safety and Immunogenicity Study of a Ross River Virus (RRV) Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Christiane Thomasser, Clinical Project Manager, Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 880701
Record Dates: First submitted 2008-07-17; First posted 2008-07-18 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Ross River Virus Disease (RRVD)
MeSH Terms: conditions — Ross River Virus Infection | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1, Treatment Arm 1 (Experimental): Randomization of a total of approx. 200 subjects to one of four treatment arms at 1:1:1:1 ratio to receive 1.25 µg of the RRV Vaccine with/without adjuvant (Al(OH)3), or 2.5 µg of the RRV Vaccine with/without adjuvant (Al(OH)3). Cohort 1 is subdivided into Cohort 1a (n = 60, i.e. 15 subjects per dose/adjuvantation combination) to receive the first vaccination on Day 0, with Day 7 safety data being reviewed by a Data Monitoring Committee and, following DMC recommendation, to receive the second vaccination at Day 21; Cohort 1b (n=140, i.e. 35 subjects per dose/adjuvantation combination) is to be vaccinated twice 21 days apart upon availability of DMC recommendation. Booster vaccination to follow 180 days after first vaccination.
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant
- Cohort 1, Treatment Arm 2 (Experimental): Same as Cohort 1, Treatment Arm 1
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant
- Cohort 1, Treatment Arm 3 (Experimental): Same as Cohort 1, Treatment Arm 1
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant
- Cohort 1, Treatment Arm 4 (Experimental): Same as Cohort 1, Treatment Arm 1
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant
- Cohort 2, Treatment Arm 1 (Experimental): Randomization of a total of approx. 100 subjects to one of two treatment arms at 1:1 ratio to receive 5 µg of the RRV Vaccine with/without adjuvant (Al(OH)3). Vaccinations take place upon review of Cohort 1a Day 7 safety data by DMC and recommendation to proceed. Booster vaccination to follow 180 days after first vaccination.
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant
- Cohort 2, Treatment Arm 2 (Experimental): Same as Cohort 2, Treatment Arm 1
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant
- Cohort 3, Treatment Arm 1 (Experimental): Randomization of a total of approx. 100 subjects to one of two treatment arms at 1:1 ratio to receive 10 µg of the RRV Vaccine with/without adjuvant (Al(OH)3). Vaccinations take place upon review of Cohort 1b and Cohort 2 Day 7 safety data by DMC and recommendation to proceed. Booster vaccination to follow 180 days after first vaccination.
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant
- Cohort 3, Treatment Arm 2 (Experimental): Same as Cohort 3, Treatment Arm 1
  Interventions: Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant

INTERVENTIONS:
Biological: Formalin-treated, UV-inactivated, whole-virion, Vero cell-derived, preservative free Ross River Virus (RRV) vaccine with or without an Al(OH)3 adjuvant — Two intramuscular injections of either 1.25 µg, 2.5 µg, 5 µg or 10 µg on Days 0 and 21, with a booster vaccination to follow 180 days after the first.

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of the Ross River Virus (RRV) Vaccine in a healthy young adult population. Other objectives of this study are to assess the immunogenicity of the RRV Vaccine in a healthy young adult population and to identify the optimal dose level of the RRV Vaccine in a healthy young adult population.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 to 40 years of age, inclusive, on the day of screening;
* Have an understanding of the study and its procedures, agree to its provisions, and give written informed consent prior to study entry;
* Are generally healthy;
* Are physically and mentally capable of participating in the study and following study procedures;
* Agree to keep a daily record of symptoms for the duration of the study;
* If female of childbearing potential - have a negative urine pregnancy test result within 24 hours of the scheduled first vaccination and agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

* Have a history of RRV exposure or a history of travel to a RRV endemic area: Australia, West Papua, Papua New Guinea, Solomon Islands, New Caledonia, Fiji Islands, Samoa Islands and Cook Island;
* Have a Body Mass Index > 35;
* Have an elevated blood pressure at screening of > 159 mmHg systolic and/or > 99 mmHg diastolic while seated and at rest and confirmed by two additional measurements taken at least 30 minutes apart (while seated and at rest);
* Have clinically significant abnormal clinical laboratory values at screening;
* Have clinically significant electrocardiographic abnormalities at screening;
* Test positive for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HbsAg) or Hepatitis C Virus (HCV);
* Have a history of cardiovascular disease;
* Have a history of immunodeficiency or autoimmune diseases;
* Have a history of arthritis (joint swelling, tenderness, warmth or erythema) on more than one occasion, not related to trauma (including running) or any episode of non-trauma related arthritis within the previous 6 months;
* Have an active neoplastic disease or have a history of hematological malignancy;
* Have a disease or are undergoing a form of treatment that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (> 800 mg/day of beclomethasone dipropionate or equivalent), corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs;
* Have a history of inflammatory or degenerative neurological disease (eg Guillain Barré, multiple sclerosis);
* Have received any vaccination within 2 weeks prior to vaccination in this study;
* Have received a blood transfusion or immunoglobulins within 30 days prior to vaccination in this study;
* Have donated blood or plasma within 30 days prior to vaccination in this study;
* Have a history of any vaccine related contraindicating event (eg, anaphylaxis, allergy to components of the test vaccine, other known contraindications);
* Have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating;
* Have a positive urine drug screen, (unless the detected drug is currently prescribed by a licensed health care provider and the continued administration of the drug would not otherwise exclude the subject from participation);
* Were administered an investigational drug within 6 weeks prior to study entry;
* Are concurrently participating in a clinical study that includes the administration of an investigational product;
* Are a member of the team conducting this study;
* Are in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study;
* If female, are pregnant or lactating.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Rates of subjects with fever with onset within 7 days after the first and 7 days after the second vaccination | Within 7 days after the first and second vaccinations
Immune response measured by RRV-specific IgG titer 21 days after the second vaccination | 21 days after the second vaccination

CONTACTS AND LOCATIONS:
Locations (10):
- Austria (2):
  - Privatklinik Leech, Graz
  - General Hospital Vienna, Department for Clinical Pharmacology, Vienna
- Belgium (2):
  - Universiteit Antwerpen VAXINFECTIO, Antwerp
  - Unité d´Investigation Clinique BioVallée, La Louvière
- Netherlands (6):
  - Andromed Breda, Breda
  - Andromed Eindhoven, Eindhoven
  - Andromed Leiden, Leiden
  - Andromed Nijmegen, Nijmegen
  - Andromed Oost, Velp
  - Andromed Zoetermeer, Zoetermeer